CLINICAL TRIAL: NCT04555213
Title: A Dose Escalation and Dose Expansion Study of NOX66 in the Treatment of COVID-19 Infection (NOXCOVID)
Brief Title: A Dose Escalation and Dose Expansion Study of NOX66 in the Treatment of COVID-19
Acronym: NOXCOVID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOX66-007
Record Dates: First submitted 2020-09-16; First posted 2020-09-18 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Part 1 Dose Escalation: 400mg, 600mg, 800mg, 1200mg & 1800mg Part 2 Dose Expansion : Recommended Phase 2 Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Cohort 1 - NOX66 400mg (Experimental): NOX66 400 mg suppository OD
  Interventions: Drug: NOX66
- Dos Escalation Cohort 2 - NOX66 600mg (Experimental): NOX66 600 mg suppository OD
  Interventions: Drug: NOX66
- Dose Escalation Cohort 3 - NOX66 800mg (Experimental): NOX66 800 mg daily (400 mg suppository BID)
  Interventions: Drug: NOX66
- Dose Escalation Cohort 4 - NOX66 1200mg (Experimental): NOX66 1200 mg daily (600 mg suppository BID)
  Interventions: Drug: NOX66
- Dose Escalation Cohort 5 - NOX66 1800mg (Experimental): NOX66 1800 mg daily (600 mg suppository TID)
  Interventions: Drug: NOX66
- Dose Expansion - NOX66 Recommended Phase 2 Dose (Experimental): Dose Expansion: NOX66 RP2D
  Interventions: Drug: NOX66

INTERVENTIONS:
Drug: NOX66 — NOX66 Suppository

SUMMARY:
Phase Ib, open-label, multicenter, study of NOX66, given rectally to hospitalized patients with moderate systemic illness due to COVID-19 infection at high risk of developing severe sepsis / septic shock.

ELIGIBILITY:
Key Inclusion Criteria:

1. Hospitalized patient with clinically diagnosis of SARS-CoV-2 virus infection per World Health Organization criteria including positive nucleic acid test of any specimen (e.g., respiratory, blood, or other bodily fluid) within 2 weeks prior to screening.{Other confirmatory test results will be accepted upon approval from Sponsor/CRO Medical Monitor prior to enrolment}.
2. Symptoms suggestive of moderate systemic illness with COVID-19, which could include any of the following symptoms: fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, or shortness of breath at rest, or respiratory distress.
3. Clinical signs indicative of moderate systemic COVID-19 illness (with high risk of developing severe ARDS/septic shock) with an aggregate of NEWS-2 score of 4-6 or 3 in one single parameter.

Key Exclusion Criteria:

Patients who meet any of the following criteria will be disqualified from entering the study:

1. Patients who require endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥ 0.5), non-invasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure.
2. Presence of any of the following abnormal laboratory values at screening: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 x upper limit of normal (ULN), platelets <50,000/µL.
3. Treatment with anti-IL 6, anti-IL-6R antagonists, or with Janus kinase inhibitors in the past 30 days or plans to receive during the study period.
4. Current treatment with conventional synthetic disease-modifying antirheumatic drugs (DMARDs)/immunosuppressive agents.
5. Use of chronic oral corticosteroids for a non-COVID-19-related condition in a dose higher than prednisone 10 mg or equivalent per day.
6. History of, or current autoimmune or inflammatory systemic or localized disease(s) other than rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 60 Days
  Routine safety monitoring during the study period

SECONDARY OUTCOMES:
Change of National Early Warning Score 2 units from baseline | 60 Days
  Measurement of 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness) to assess overall clinical condition.
Change in WHO-9 point ordinal scale | 60 Days
  Assessment of WHO-9 point ordinal scale for clinical improvement (i.e., 0 = uninfected and 8 = death) category ordinal scale of clinical status from admission.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Mautner, MD, PhD, Study Director — Noxopharm Limited
Locations (1):
- Institute of Emergency Medicine, Chisinau, Moldova